CLINICAL TRIAL: NCT06911255
Title: A Phase I/IIa, Single-arm, Open-label, IIT for Safety and Efficacy Evaluation of Tremelimumab Plus Durvalumab(MEDI4736) in Combination With Concurrent Transarterial Chemoembolization in Unresectable Hepatocellular Carcinoma
Brief Title: Safety and Efficacy of Tremelimumab+Durvalumab(MEDI4736)+TACE in Unresectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yoon Jun Kim (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Yoon Jun Kim, Coordinating Investigator, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DETECT
Record Dates: First submitted 2025-01-08; First posted 2025-04-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma (HCC); Unresectable Hepatocellular Carcinoma
Keywords: HCC Durvalumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Intervention Model Description: After the intravenous (IV) administration of 300 mg of tremelimumab and 1,500 mg of durvalumab, transarterial chemoembolization (TACE) will be performed in combination with 1,500 mg of durvalumab via IV infusion every 4 weeks (Q4W) until disease progression (PD) is confirmed. TACE will be carried out 1 to 2 weeks (7 to 14 days) after the administration of tremelimumab + durvalumab, and thereafter, it will be performed as needed at the discretion of the investigator during the treatment period. If additional TACE is performed, there must be at least a 1-week interval between the additional TACE and the administration of durvalumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tremelimumab Plus Durvalumab (MEDI4736) in Combination with Concurrent Transarterial Chemoembolizati (Experimental): After the intravenous (IV) administration of 300 mg of tremelimumab and 1,500 mg of durvalumab, transarterial chemoembolization (TACE) will be performed in combination with 1,500 mg of durvalumab via IV infusion every 4 weeks (Q4W) until disease progression (PD) is confirmed. TACE will be carried out 1 to 2 weeks (7 to 14 days) after the administration of tremelimumab + durvalumab, and thereafter, it will be performed as needed at the discretion of the investigator during the treatment period. If additional TACE is performed, there must be at least a 1-week interval between the additional TACE and the administration of durvalumab.
  Interventions: Drug: Tremelimumab Plus Durvalumab (MEDI4736); Procedure: Transarterial chemoembolization (TACE)

INTERVENTIONS:
Drug: Tremelimumab Plus Durvalumab (MEDI4736) — Study subjects will receive 1,500 mg of durvalumab intravenously every 4 weeks until PD is observed. However, treatment will be discontinued if unacceptable toxicity, withdrawal of consent, or any other discontinuation criteria are met. Tremelimumab will be administered first, and durvalumab infusion will begin approximately 1 hour (up to 2 hours) after the completion of tremelimumab infusion. The standard infusion time for each drug is 1 hour, but if the infusion is temporarily interrupted, the total duration should not exceed 8 hours at room temperature.
  Other Names: Imfinzi®; Imjudo
Procedure: Transarterial chemoembolization (TACE) — TACE will be carried out 1 to 2 weeks (7 to 14 days) after the administration of tremelimumab + durvalumab, and thereafter, it will be performed as needed at the discretion of the investigator during the treatment period. If additional TACE is performed, there must be at least a 1-week interval between the additional TACE and the administration of durvalumab.

SUMMARY:
Safety and Efficacy Evaluation of Tremelimumab Plus Durvalumab(MEDI4736) in Combination with Concurrent Transarterial Chemoembolization in Unresectable Hepatocellular carcinoma

DETAILED DESCRIPTION:
The purpose of this clinical trial is to evaluate the safety and efficacy of tremelimumab + durvalumab administered concurrently with transarterial chemoembolization (TACE) in patients diagnosed with hepatocellular carcinoma (HCC) who are not eligible for curative liver resection.

Primary Objective:

The primary objective of this clinical trial is to evaluate progression-free survival (PFS) from the time of registration using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

Secondary Objectives:

Overall Survival (OS):

To assess the overall survival from the first dose of the study drug until the data cutoff point, as determined by the investigator.

Objective Response Rate (ORR):

To assess the objective response rate of target and non-target lesions using mRECIST and RECIST 1.1. Evaluations will occur every 8 weeks after 12 weeks and for the first 48 weeks from the time of registration, and then every 12 weeks thereafter.

Time to Progression (TTP):

To measure the time from registration to disease progression using mRECIST and RECIST 1.1.

Safety Evaluation:

To evaluate the safety of tremelimumab and durvalumab, including adverse events, vital signs (blood pressure and pulse rate), and laboratory safety assessments (clinical chemistry, hematology, etc.), by assessing changes from baseline.

ELIGIBILITY:
Inclusion Criteria:

* 1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.

  2. Male or female, aged ≥19 years at time of study entry. 3. Diagnosed with unequivocal HCC confirmed histologically or diagnosed radiologically according to American Association for the Study of Liver Diseases practice guideline.

  4. Barcelona clinic liver cancer (BCLC) staging intermediate (B) stage or BCLC advanced stage (C) HCC with or without minimal extrahepatic disease (single-organ metastasis, ≤5 metastatic lesions).

  5. Must have at least 1 untreated measurable disease (untreated target lesion i.e. a viable lesion that has never been treated with locoregional treatment [transarterial chemoembolization {TACE}, TARE, percutaneous ethanol injection therapy, or radiofrequency ablation]).

  6. Child-Pugh score 5 or 6 points (Child-Pugh class A). 7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 8. Life expectancy of ≥ 12 weeks. 9. Body weight >30 kg. 10. Adequate normal organ and marrow function as defined below:
* Hemoglobin ≥9.0 g/dL
* Absolute neutrophil count (ANC) ≥1500 per mm3
* Platelet count ≥75,000 per mm3
* Albumin ≥2.8 g/dL
* Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). (This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with the Investigator).
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤5 x institutional ULN
* Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24- hour urine collection for determination of creatinine clearance:

Males:

Creatinine CL (mL/min) Females:

Creatinine CL (mL/min)

* Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)
* Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL) 11. Female patients must be either postmenopausal or, if premenopausal, must have a negative pregnancy test and agree to use 2 forms of contraception, if sexually active during their study participation.

Male patients must be surgically sterile or, if sexually active and having a pre-menopausal female partner then, must be using an acceptable form of contraception.

Adequate contraception allowed in this trial is as follows:

* Hormonal contraceptives such as combined oral contraceptive pill
* Intrauterine devices or the implantation of intrauterine system (IUS)
* Blockage methods (spermicides and condoms/spermicides and vaginal diaphragm for contraception, vaginal sponges or cervical cap) • Blockage methods (spermicides and condoms/spermicides and vaginal diaphragm for contraception, vaginal sponges or cervical cap)
* Sterilization surgery such as tubal ligation in females and vasectomy in males. 12. Evidence of postmenopausal status or negative urinary or serum pregnancy test for female premenopausal patients. Women will be considered postmenopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:
* Women <50 years of age would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the postmenopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
* Women ≥50 years of age would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

  13. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* 1. Eligible for potentially curative treatment (surgical resection, radiofrequency ablation or immediate liver transplantation).

  2. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti- Cytotoxic T-lymphocyte- associated antigen-4 (anti-CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune pathways, including prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.

  3. History of organ transplantation or hematopoietic stem cell transplantation.

  4. Any other concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, papillary thyroid cancer, early gastric cancer, or other cancer for which the patient has been disease-free for at least five years.

  5. A history of a severe contrast allergy (i.e. anaphylaxis) not controlled with premedication.

  6. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the investigational product (IP) or interpretation of patient safety or study results.

  7. Participation in another clinical study with an IP during the last 8 weeks or 5 half-lives of the study drug, whichever is longer, prior to screening.

  8. Concurrent enrolment in another clinical study, unless it is an observational (non- interventional) clinical study or during the follow-up period of an interventional study.

  9. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤1 cycle length or 14 days, whichever is longer, prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as determined by the Investigator.

  10. Any unresolved toxicity NCI-CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
* Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab and/or tremelimumab may be included at the discretion of the Investigator.

  11. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

  12. Prior hepatic radiation therapy including Total Body Irradiation (TBI) for HCC or other malignancy.

  13. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.

  14. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:
* Patients with vitiligo or alopecia
* Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Patients without active disease in the last 5 years may be included but only after consultation with the study physician
* Patients with celiac disease controlled by diet alone 15. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent.

  16. History of leptomeningeal carcinomatosis. 17. History of active primary immunodeficiency, including known positive tests for human immunodeficiency virus (HIV 1/2 antibodies).

  18. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), other than chronic infection of HBV or HCV. Participants with chronic HBV infection (positive hepatitis B surface antigen [HBsAg] and/or detectable HBV DNA) are eligible if they are receiving nucleos(t)ide analog treatment, as determined by the physician's judgment and in accordance with local practice guidelines. Those with a past or resolved HBV infection (defined as the presence of anti-hepatitis B core antibody and absence of HBsAg) are also eligible. For chronic HCV infection, participants positive for HCV antibody are eligible only if polymerase chain reaction for HCV RNA is negative.

  19. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab and/or tremelimumab. The following are exceptions to this criterion:
* Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
* Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., Computed tomography [CT] scan premedication) 20. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.

Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.

21. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth from screening to 90 days after the last dose of durvalumab and/or tremelimumab, or 180 days after the last TACE.

22. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

23. Judgment by the Investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | the time from the first study treatment administration until the date of objective disease progression
  The primary endpoint for evaluating progression-free survival (PFS) will be assessed through RECIST 1.1 evaluation.

SECONDARY OUTCOMES:
OS | the time from the first study treatment administration until death due to any cause, regardless of whether the patient withdraws from therapy or receives another anticancer therapy.
  Overall Survival (OS) from first dose of study drug until the time of data cut-off, as determined by the Investigator.
ORR | From date of enrollment until the date of first documented progression, assessed every 8 weeks up to 12 months.
  Objective Response Rate (ORR) of Target Lesion(s) and Non-Target Lesion(s)
TTP | the time from the first study treatment administration until the first confirmed tumor progression (PD) based on the RECIST 1.1 assessment.
  Time to progression (TTP) of enrollment to disease progression as assessed by RECIST 1.1 and mRECIST.
Safety of durvalumab and tremelimumab in terms of the occurrence of adverse events | Until 30 days after TACE or the last dose of tremelimumab and/or durvalumab
  changes from baseline in vital signs (blood pressure and heart rate), and safety laboratory findings (chemistry, hematology, and so on)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Jun Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No